CLINICAL TRIAL: NCT03943394
Title: PCM1-JAK2 Fusion Gene Detection in Patients With Therapy Related Myelodysplastic Syndrome / Acute Myeloid Leukemia Patients
Brief Title: PCM1-JAK2 in Therapy Related Neoplasms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RHNAhmed, assistant lecturer, Assiut University
Other Study IDs: PCM1-JAK2 fusion gene
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Detection of PCM1-JAK2 Fusion Gene by FISH in the Two Types of t-MDS/AML and Relationship Between PCM1-JAK2 Fusion Gene and Cumulative Dose, Dose Intensity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Denovo MDS/ AML: Patients with de-novo myeloid neoplasm either myelodysplastic syndrome and/ or acute myeloid leukemia which are diagnosed by complete blood count , blood film, bone marrow aspirate, bone marrow biopsy , immunophenotyping and bone marrow biopsy with these inclusion criteria • Myelodysplastic syndromes: the diagnosis of MDS must be confirmed by a bone marrow aspirate and/or biopsy : blast count must be < 20%;
  • Acute myeloid leukemia with multilineage dysplasia: the diagnosis of AML-TLD must be confirmed by a bone marrow aspirate and/or biopsy NOTE: there must be evidence of >= 20% blasts on the review of the bone marrow aspirate and/or biopsy;
  Interventions: Other: fresh samples are obtained from patients for detction of PCM1- JAK2 fusion gene
- therapy related MDS/ AML: PCM1-JAK2 fusion gene detection in patients with therapy related Myelodysplastic syndrome / Acute myeloid leukemia patients
  Interventions: Other: fresh samples are obtained from patients for detction of PCM1- JAK2 fusion gene

INTERVENTIONS:
Other: fresh samples are obtained from patients for detction of PCM1- JAK2 fusion gene — Samples are dehydrated in ethanol (a 50, 80 and 95% (v/v) series, exposure for 3 min to 300 µl ethanol at each concentration) prior to hybridization.
  Samples on tapes are hybridized for 15 minutes at 55?C using a moisture-sealed slide incubation chamber. Briefly, 500 µl volumes of hybridization buffer (0.7 M NaCl, 0.1 M Tris [pH 8.0], 0.1% sodium dodecyl sulfate, 10 mM EDTA, containing probe, preheated to 55 ºC) are applied to the surface of the tape and the chamber's lid is sealed, creating a moist, temperature controlled environment within the chamber.
  After 15 min, the lid is removed and samples are briefly rinsed with probe-free hybridization buffer, preheated to 55ºC.
  Hybridized cells on tapes are counterstained for 10 minutes in the dark with ~30 µl mounting medium containing 1.5 µg ml-1 4',6-diamidino-2-phenylindole (DAPI).
  Then tapes are mounted with a coverslip and examined using a fluorescence microscope.

SUMMARY:
The term "therapy-related" leukemia is descriptive and is based on a patient's history of exposure to cytotoxic agents. Although a causal relationship is implied, the mechanism remains to be proven. These neoplasms are thought to be the direct consequence of mutational events induced by the prior therapy Therapy-related myelodysplastic syndromes / acute myeloid leukemia (t- MDS / t-AML) is now considered a single entity, called therapy-related myeloid neoplasms based on the current World Health Organization WHO classification2,. It is a well-recognized clinical syndrome occurring as a late complication following Cytotoxic agents and ionizing radiotherapy in the treatment of most cancer types: Hodgkin lymphoma (HL), non-Hodgkin lymphoma (NHL), acute lymphoblastic leukemia (ALL), sarcoma, and ovarian and testicular cancerThe incidence of t-MDS/AML following conventional therapy ranges from 0.8% to 6.3% at 20 years. The median time to development of t-MDS/AML is 3 to 5 years, with the risk decreasing markedly after the first decade Two types of t-MDS/AML are recognized in the WHO classification depending on the causative therapeutic exposure: an alkylating agent/radiation-related type and a topoisomerase II inhibitor-related type. Alkylating agent-related t-MDS/AML usually appears 4 to 7 years after exposure to the mutagenic agent .The reciprocal translocation t(8;9) (p22;p24) between the short arm of chromosome 8 and the long arm of chromosome 9 is a recurrent abnormality that fuses the Janus activated kinase 2 (JAK2) to the human autoantigen pericentriolar material 1 gene (PCM1) , with breakage and reunion at bands 8p11 and 9q3410Due to PCM1-JAK2 gene fusion, the coiled-coil domains of PCM1 mediate an oligomerization that brings together the linked JAK2 domains resulting in a constitutively activated tyrosine kinase domain of JAK2The most common mechanism for JAK2 activation in hematologic malignancies is the point mutation at position 617 (V617F).

The consequences of JAK2 activation are neoplastic transformation and abnormal cell proliferation in various malignancies

* So, translocations involving the JAK2 locus are considered of oncogenic importance in acute leukemias and myelodysplastic/ myeloproliferative diseases.
* Patients with this abnormality present with broad clinical spectrum ranging from chronic to acute hematological diseases with myeloid or lymphoid appearance

DETAILED DESCRIPTION:
The term "therapy-related" leukemia is descriptive and is based on a patient's history of exposure to cytotoxic agents. Although a causal relationship is implied, the mechanism remains to be proven. These neoplasms are thought to be the direct consequence of mutational events induced by the prior therapy .

Therapy-related myelodysplastic syndromes / acute myeloid leukemia (t- MDS / t-AML) is now considered a single entity, called therapy-related myeloid neoplasms based on the current World Health Organization WHO classification2,. It is a well-recognized clinical syndrome occurring as a late complication following Cytotoxic agents and ionizing radiotherapy in the treatment of most cancer types: Hodgkin lymphoma (HL), non-Hodgkin lymphoma (NHL), acute lymphoblastic leukemia (ALL), sarcoma, and ovarian and testicular cancer3,4.

The characteristics of therapy-related myeloid neoplasm and the timing of its development after a primary diagnosis depend on the exposure to specific agents as well as the cumulative dose and dose intensity of the preceding cytotoxic therapy 5.

The incidence of t-MDS/AML following conventional therapy ranges from 0.8% to 6.3% at 20 years. The median time to development of t-MDS/AML is 3 to 5 years, with the risk decreasing markedly after the first decade 6.

Two types of t-MDS/AML are recognized in the WHO classification depending on the causative therapeutic exposure: an alkylating agent/radiation-related type and a topoisomerase II inhibitor-related type. Alkylating agent-related t-MDS/AML usually appears 4 to 7 years after exposure to the mutagenic agent .

Approximately two-thirds of patients present with MDS and the remainder with AML with myelodysplastic features. Patients frequently present with cytopenias. Multilineage dysplasia is often present 7.

In this classic form of therapy-related leukemia that follows treatment with alkylating agents and/or radiation therapy, the blood and bone marrow findings resemble those seen in primary MDS, although the degree of dysgranulopoiesis and dysmegakaryocytopoiesis is typically greater 8.

In contrast to alkylating agent t-MDS/AML, AML secondary to topoisomerase II inhibitors often does not have a preceding myelodysplastic phase, and presents as overt acute leukemia, often with a prominent monocytic component. The latency period between the initiation of treatment with topoisomerase II inhibitors and the onset of leukemia is brief, with a median of 2 to 3 years 9.

The reciprocal translocation t(8;9) (p22;p24) between the short arm of chromosome 8 and the long arm of chromosome 9 is a recurrent abnormality that fuses the Janus activated kinase 2 (JAK2) to the human autoantigen pericentriolar material 1 gene (PCM1) , with breakage and reunion at bands 8p11 and 9q341010.

PCM1 encodes a large protein of 228kDa containing several potential coiled-coil domains in its aminoterminal part. This protein is localized in cytoplasmatic granules referred to as centriolar satellites. It is supposed to play a crucial role in the assembly of centrosomal proteins, microtubule organisation, and in the progression of cell cycle11.

Due to PCM1-JAK2 gene fusion, the coiled-coil domains of PCM1 mediate an oligomerization that brings together the linked JAK2 domains resulting in a constitutively activated tyrosine kinase domain of JAK212, 13.

JAK2 is a member of the Janus family of tyrosine kinases (JAK1, JAK2, JAK3, TYK2). These non-receptor tyrosine kinases play a significant role in various signal transduction pathways that regulate cellular survival, proliferation, differentiation, and apoptosis. The protein is formed of seven domains. The JH2 domain (pseudokinase domain, kinase-like domain) is located in exon 14 and has an essential negative autoregulatory function14.

The most common mechanism for JAK2 activation in hematologic malignancies is the point mutation at position 617 (V617F).

The consequences of JAK2 activation are neoplastic transformation and abnormal cell proliferation in various malignancies15.

* So, translocations involving the JAK2 locus are considered of oncogenic importance in acute leukemias and myelodysplastic/ myeloproliferative diseases.
* Patients with this abnormality present with broad clinical spectrum ranging from chronic to acute hematological diseases with myeloid or lymphoid appearance 16.

Fluorescence in situ hybridization (FISH) is a kind of cytogenetic technique that allows the visualization of defined nucleic acid sequences in particular cellular or chromosomal sites by hybridization of complementary fluorescently labeled probe sequences within intact metaphase or interphase cells.

The fluorescent probes are nucleic acid labeled with fluorescent groups and can bind to specific DNA/RNA sequences. Fluorescence microscopy can be used to find out where the fluorescent probe is bound to the chromosomes17.

ELIGIBILITY:
Inclusion Criteria:

* • Myelodysplastic syndromes: the diagnosis of MDS must be confirmed by a bone marrow aspirate and/or biopsy : blast count must be < 20%; patients with any International Prognostic Score (IPSS) are eligible; patients with low or intermediate (INT)-1 IPSS must have a platelet count < 50x10⁹/L and/or absolute neutrophil count (ANC) < 50x10⁹/L.

  * Acute myeloid leukemia with multilineage dysplasia: the diagnosis of AML-TLD must be confirmed by a bone marrow aspirate and/or biopsy NOTE: there must be evidence of >= 20% blasts on the review of the bone marrow aspirate and/or biopsy; AML-TLD will be interpreted to include patients formerly diagnosed by French-American-British (FAB) criteria as refractory anemia with excess blasts in transformation (RAEB-t), as well as patients with no history of antecedent hematologic disorder who have AML which meets criteria for AML-TLD by World Health Organization (WHO) criteria; patients with AML-TLD must have a white blood cell (WBC) =< 30x10⁹/L documented within 4 weeks prior to study entry (two sets of counts that are 2 weeks apart will be taken); patients whose WBC has doubled within this period of time and is greater than 20x10⁹/L at the time of screening will not be eligible
  * Patients have started therapy (cytotoxic agents and ionizing radiotherapy) at least 2 years ago.

Exclusion Criteria:

* other therapy related neoplasms other than myelodplastic syndrome or acute myeloid leukemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: therapy related acute myeloid leukemia and / or myelodysplastic syndrome
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Detection of PCM1-JAK2fusion gene | 24 months
  Using fresh sample from patients with myeloid neoplasm to search for PCM1-JAK2 fusion gene in the 2 types of thaerap related myeloid neoplasm , studying relationship between PCM1-JAK2 and dose intensity and time of exposure, and studying relationship between PCM1-JAK2 and other cytogenetic abnormalities by using FISH technique and

IPD SHARING:
Plan to Share IPD: No